CLINICAL TRIAL: NCT01595633
Title: Randomized Study Comparing Nucleoside Analogues Plus Tenofovir and Nucleoside Analogues Plus Adefovir in Chronic Hepatitis B Patients With Suboptimal Response to Adefovir-based Combination Therapy Due to Nucleoside Analogues Resistance
Brief Title: Switch From Adefovir to Tenofovir in Chronic Hepatitis B for Suboptimal Response to Adefovir-based Combination Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sang Hoon Ahn, Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0937
Record Dates: First submitted 2012-03-11; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis B
Keywords: nucleoside analogue; adefovir; tenofovir; hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adefovir, nucleoside analogues (Active Comparator): Nucleoside analogues (Lamivudine 100mg, Telbivudine 600mg, Entecavir 1mg, or Clevudine 30mg) + Adefovir 10mg
  Interventions: Drug: Switching from adefovir (10mg/day) to tenofovir (300mg/day)
- Tenofovir, nucleoside analogues (Experimental): Nucleoside analogues (Lamivudine 100mg, Telbivudine 600mg, Entecavir 1mg, or Clevudine 30mg) + Tenofovir 300mg
  Interventions: Drug: Switching from adefovir (10mg/day) to tenofovir (300mg/day)

INTERVENTIONS:
Drug: Switching from adefovir (10mg/day) to tenofovir (300mg/day) — active comparator: Nucleoside analogues (Lamivudine 100mg, Telbivudine 600mg, Entecavir 1mg, or Clevudine 30mg/day) + Adefovir 10mg/day Experimental: Nucleoside analogues (Lamivudine 100mg, Telbivudine 600mg, Entecavir 1mg, or Clevudine 30mg/day) + Tenofovir 300mg/day

SUMMARY:
In Korea, the number of suboptimal responders to rescue combination therapy is also increasing. As a matter of fact, according to the investigations in Korea, HBV DNA undetectability at 48 weeks of adefovir and lamivudine combination rescue therapy for patients with lamivudine resistance was reported to be only 32.4%, which suggested that the appropriate another rescue therapy might be urgently required. However, there is no promising oral antiviral agents to control these patients in Asia-Pacific region, where tenofovir is not widely available. Tenofovir has a higher potent antiviral efficacy and a negligible drug resistance rate. The switch from adefovir to tenofovir in patients who have insufficient hepatitis B virus (HBV) suppression (HBV DNA ≥ 60 IU/mL by PCR) may lead to increased viral suppression or more HBeAg loss/seroconversion.

Here, the investigators aimed to conduct a randomized study on evaluating the antiviral efficacy, safety, and tolerability of switching from adefovir to tenofovir in chronic hepatitis B patients who have suboptimal response to adefovir-based combination rescue therapy due to nucleoside analogues Resistance (SATIS study).

DETAILED DESCRIPTION:
The major goal of antiviral therapy against chronic hepatitis B is to suppress viral replications successfully, ultimately preventing the chronic liver damage, development of liver cirrhosis and hepatocellular carcinoma. In Korea, the number of multi-drug resistant CHB has been rapidly increased last few years. It is because that the national health insurance coverage is very limited for the patients who experienced primary treatment failure. The only switch to adefovir has been allowed in lamivudine resistant patients and thus this sequential rescue therapy generated multi-drug resistance to both adefovir and another drugs. Thus, nowadays, add-on therapy rather than switch therapy might be preferred from major guidelines in this point.

However, the number of suboptimal responders to rescue combination therapy is also increasing. As a matter of fact, according to the investigations in Korea, HBV DNA undetectability at 48 weeks of adefovir and lamivudine combination rescue therapy for patients with lamivudine resistance was reported to be only 32.4%, which suggested that the appropriate another rescue therapy might be urgently required. However, there is no promising oral antiviral agents to control these patients in Asia-Pacific region, where tenofovir is not widely available. Tenofovir has a higher potent antiviral efficacy and a negligible drug resistance rate. It belongs to the different class compared to other oral nucleoside analogues (NAs) such as lamivudine, telbivudine, clevudine and entecavir. The switch from adefovir to tenofovir in patients who have insufficient hepatitis B virus (HBV) suppression (HBV DNA ≥ 60 IU/mL by PCR) may lead to increased viral suppression or more HBeAg loss/seroconversion. The results of this study will provide a rationale for switch from adefovir to tenofovir in combination to another drug continued (lamivudine, telbivudine, clevudine and entecavir).

Here, the investigators aimed to conduct a randomized study on evaluating the antiviral efficacy, safety, and tolerability of switching from adefovir to tenofovir in chronic hepatitis B patients who have suboptimal response to adefovir-based combination rescue therapy due to nucleoside analogues Resistance (SATIS study).

ELIGIBILITY:
Inclusion Criteria:

* subjects with age >= 20 years
* subjects with chronic hepatitis B
* subjects treated with nucleoside analogues plus adefovir for at least 6 months due to resistance to nucleoside analogues (Lamivudine, Telbivudine, Entecavir, or Clevudine)
* subjects with partial virologic response to nucleoside analogues plus adefovir HBV DNA ≥ 60 IU/mL)
* subjects with ALT less than 5 times of upper limit of normal
* subjects who agreed to participate in the clinical trials and signed the informed consents

Exclusion Criteria:

* subjects with decompensate liver cirrhosis Child-Pugh B, C)
* subjects with Adefovir mutation
* subjects with HCV, HDV, or HIV infection
* pregnant or lactating women
* women of childbearing age who do not use the appropriate contraception method
* subjects who have the abnormal lesion suspected of hepatocellular carcinoma on imaging modalities
* subjects with other liver diseases such as hemochromatosis, Wilson's disease, alcoholic liver disease, nonalcoholic liver disease, alpha-1 antitrypsin deficiency
* subjects with hypersensitivity for study drugs
* subjects who participated in other clinical trials 60 days before the current recruitment
* subjects who are judged as inappropriate by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
number of patients with complete virologic response (HBV DNA < 60 IU/mL, approximately 300 copies/mL) at 48 weeks treatment | 48 weeks
  Complete virologic response (HBV DNA < 60 IU/mL, approximately 300 copies/mL) at 48 weeks treatment

SECONDARY OUTCOMES:
number of patients with antiviral response at 48 weeks therapy | 48 weeks
  number of patients with antiviral response (defined as decrement of HBV DNA level with 2 Log from baseline) at 48 weeks therapy
number of patients with biochemical response at 48 weeks therapy | 48 weeks
  number of patients with biochemical response (defined as ALT normalization) at 48 weeks therapy
number of patients with serologic response at 48 weeks therapy | 48 weeks
  number of patients with serologic response (defined as HBeAg seroconversion in case of HBeAg-positive hepatitis) at 48 weeks therapy
number of patients with appearance of resistant mutant strain at 48 weeks | 48 weeks
  number of patients with appearance of resistant mutant strain at 48 weeks
Number of Participants with Adverse Events | 48 weeks
  Number of Participants with Adverse Events during treatments (Adverse effects will be monitored every visit using physical examination and routine blood chemistry tests.)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, MD, PhD., Principal Investigator — Department of Internal Medicine, Yonsei University College of Medicine
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea